CLINICAL TRIAL: NCT03087448
Title: A Phase I/II Study of Ceritinib + Trametinib in Patients With Advanced ALK-Positive Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Ceritinib + Trametinib in Patients With Advanced ALK-Positive Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis Pharmaceuticals (Industry); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 166512; NCI-2017-01318 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-02-10; First posted 2017-03-22 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ALK rearranged; Stage IIIB NSCLC; Stage IV NSCLC; ROS-1 rearranged NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ceritinib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ceritinib + Trametinib (Experimental): PHASE 1 Standard 3+3 dose escalation starting at dose level 1. Patients with ALK-rearranged, or ROS-1 rearranged NSCLC. 6-18 patients will be enrolled.
  Ceritinib dose: 300-450mg orally, once daily over 28 day cycles. Trametinib dose: 1.5mg-2.0mg orally, once daily over 28 day cycles.
  PHASE II The study was terminated before Phase II was initiated. The study did not open Phase II for enrollment.
  Interventions: Drug: Ceritinib; Drug: Trametinib

INTERVENTIONS:
Drug: Ceritinib — ALK tyrosine inhibitor, 300 mg - 450 mg PO daily.
  Phase I dose escalation:
  1. Ceritinib 300mg
  2. Ceritinib 450mg
  3. Ceritinib 450mg
  The Phase II doses will be determined by Phase I dose escalation study
  Other Names: Zykadia
Drug: Trametinib — MEK kinase inhibitor, 1.5 mg - 2.0 mg PO daily.
  Phase I dose escalation:
  1. Trametinib 1.5mg
  2. Trametinib 1.5mg
  3. Trametinib 2.0mg
  The Phase II doses will be determined by Phase I dose escalation study
  Other Names: Mekinist

SUMMARY:
This is a phase I/II study of ceritinib and trametinib in Stage IIIB or IV anaplastic lymphoma kinase (ALK) rearranged non-small cell lung cancer (NSCLC). The Phase I portion will investigate the safety and tolerability of the combination of ceritinib and trametinib in ALK or ROS-1 rearranged NSCLC. The Phase II portion will investigate the clinical efficiency of the combination of ceritinib and trametinib in 3 single arm cohorts: ALKi (ALK inhibitor) naïve patients; post-crizotinib progressed disease (PD) patients; and PD second line ALK tyrosine kinase inhibitor (TKI) patients.

DETAILED DESCRIPTION:
This was intended to be a phase I/II study of ceritinib and trametinib in Stage IIIB or IV ALK rearranged NSCLC.

The phase I portion is a standard 3+3 dose escalation study starting at dose level 1 and will be open to any patient with ALK-rearranged, or ROS-1 rearranged NSCLC.

The study was terminated before Phase II was initiated. The study did not open Phase II for enrollment into the planned cohorts:

* Cohort A (ALKi Naïve)
* Cohort B (Post-crizotinib PD)
* Cohort C (PD second line ALK TKI (e.g., alectinib, ceritinib, PF-06463922 or - AP21163)

Only participants in Phase 1 were enrolled.

Patients may continue treatment for up to 24 months from the time of study entry, and will receive 12 months of follow-up following completion of the drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or older.
2. Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
3. Women of childbearing potential must have a negative serum pregnancy test within 3 days prior to Cycle 1 Day 1 and agree to use effective contraception, throughout the treatment period, and for 4 months after the last dose of study treatment.

   .
4. Patients must have histologically or cytological confirmed stage IIIB or IV non-small cell lung cancer.
5. Documented ALK-rearrangement (or ROS1 rearrangement for phase I only) break-apart fluorescence in situ hybridization (FISH) (in at least 15% of tumor cells), or next generation sequencing assay performed on tumor sample or cell-free DNA in Clinical Laboratory Improvement Amendments (CLIA)-approved laboratory.
6. Measurable disease defined by RECIST 1.1 criteria
7. Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2.
8. Life expectancy of at least 3 months.
9. Resolution of all acute toxic effects of prior chemotherapy, immunotherapy, radiotherapy or surgical procedures to ≤ grade 2 (CTCAE v 4.0). Exception to this criterion: patients with any grade of alopecia are allowed to enter the treatment.
10. The following laboratory criteria have been met:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Hemoglobin (Hgb) ≥ 9 g/dL
    * Platelets ≥ 75 x 109/L
    * Prothrombin time (PT) / international normalized ratio (INR) and Partial thromboplastin time (PTT) ≤1.5 x upper limit of normal (ULN)
    * Serum creatinine ≤ 1.5 mg/dL and /or calculated creatinine clearance (using Cockcroft-Gault formula) ≥ 30 mL/min
    * Albumin 2.5 g/dL
    * Total bilirubin ≤ 1.5 x ULN, except for patients with Gilbert's syndrome who may be included if total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
    * Aspartate transaminase (AST) ≤ 2.5 x ULN; alanine transaminase (ALT) ≤ 2.5 x ULN, except for patients with liver metastasis, who are only included if AST and ALT < 5 x ULN
    * Alkaline phosphatase (ALP) ≤ 5.0 x ULN
    * Fasting plasma glucose ≤ 175 mg/dL (≤ 9.8 mmol/L)
    * Serum amylase ≤ 2 x ULN
    * Serum lipase ≤ ULN
11. Patient must have the following laboratory values or have the following laboratory values corrected with supplements to be within normal limits before the first dose of ceritinib + trametinib:

    * Potassium
    * Magnesium
    * Phosphorus
    * Total calcium (corrected for serum albumin)
12. Left Ventricular Ejection fraction (LVEF) ≥ lower limit of normal (LLN) by echocardiogram (ECHO) or multigated acquisition scan (MUGA)
13. Patient has the ability to understand and provide signed informed consent.
14. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedure.
15. Specific inclusion criteria for the phase II dose expansion cohorts:

Documented ALK-rearranged stage IIIB or IV NSCLC and:

* Cohort A: No prior ALK inhibitor therapy (prior chemotherapy or immunotherapy is allowed).
* Cohort B: Prior treatment with crizotinib and documented disease progression by RECIST 1.1 criteria.
* Cohort C: Prior treatment with 2nd generation ALKi (e.g. ceritinib, alectinib, loratinib, or brigatinib) and documented disease progression by RECIST 1.1 criteria.

Exclusion Criteria:

1. Patients with known hypersensitivity to any of the excipients of ceritinib (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate).
2. Patient has history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).
3. Patient who has received thoracic radiotherapy to lung fields ≤4 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs) radiotherapy ≤2 weeks prior to starting the study treatment or has not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤2 weeks prior to starting study treatment is allowed.
4. Prior systemic anti-cancer treatment (chemotherapy, immunotherapy, biologic therapy, vaccine therapy, or investigational treatment) within the last 3 weeks, or chemotherapy without delayed toxicity within the last 2 weeks preceding the first dose of the combination. Prior systemic treatment in the adjuvant setting is allowed.
5. Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:

   * unstable angina within 6 months prior to screening;
   * myocardial infarction within 6 months prior to screening;
   * history of documented congestive heart failure (New York Heart Association functional classification III-IV);
   * Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication
   * initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;
   * ventricular arrhythmias
   * supraventricular and nodal arrhythmias not controlled with medication;
   * other cardiac arrhythmia not controlled with medication;
   * corrected QT (QTcF) > 470 ms using Fridericia's correction on the screening electrocardiogram (ECG)
6. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of orally administered medication (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
7. Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with ceritinib and for the duration of participation:

   * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (please refer to http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm)
   * Strong inhibitors or strong inducers of CYP3A4/5 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
   * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, and/or CYP2C9 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
   * Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed (eg, dabigatran, rivaroxaban, apixaban).
   * Unstable or increasing doses of corticosteroids; If patients are on corticosteroids for endocrine deficiencies or tumor-associated symptoms, dose must have been stabilized (or decreasing) for at least 5 days before first dose of study treatment.
   * Enzyme-inducing anticonvulsive agents
   * Herbal supplements
8. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human Chorionic Gonadotropin (hCG) laboratory test.
9. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months after the last dose of study treatment. Highly effective contraception methods include:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization (at least 6 months prior to screening) with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
   * Combination of any two of the following (a+b or a+c or b+c):

     1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
     3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

   In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

   Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile. (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
10. Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after the last dose of study treatment. Male patients for 3 months should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
11. Patient has a history of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease.
12. Patient has other severe, acute, or chronic medical conditions including uncontrolled diabetes mellitus or psychiatric conditions or laboratory abnormalities that, in the opinion of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
13. Patient has had major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior to starting study treatment or has not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can receive study treatment ≥ 1 week after these procedures.
14. History of another malignancy. Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer and/or subjects with indolent (early stage breast cancer or prostate cancer) second malignancies are eligible after discussion with the study principle investigator (PI).
15. History of retinal vein occlusion (RVO)
16. Symptomatic brain metastases or leptomeningeal (LM) disease requiring corticosteroids for symptom management. Asymptomatic brain metastases or LM will be allowed on study.
17. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 12 weeks.
  Determine the maximum tolerated dose (MTD) by evaluating the number and frequency of Adverse Events (AEs) as determined by National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0 by investigator assessment, and identify a recommended phase II dose (RP2D) for phase II dose expansion cohorts.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 1 year
  The ORR is defined as the best overall response recorded from the start of the treatment until disease progression or recurrence as assessed over a 1-year period from the start of treatment. The percentages of patients with a best overall response rate of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be determined.
Disease control rate (DCR) | Up to 1 year
  DCR will be defined as the percentage of patients who have achieved CR, PR, or SD for at least 12 weeks
Median Progression-free survival (PFS) | Up to 2 years
  PFS will be calculated as 1+ the number of days from the first dose of study drugs to documented radiographic progression or death due to any cause over a period of 18 months. For patients who continue treatment post-progression, the date of radiographic progression will be used for PFS analysis. The Kaplan-Meier analysis will be used to calculate the mean PFS with 95% confidence interval.
Median Overall survival (OS) | Up to 18 months
  OS will be calculated as 1+ the number of days from the first dose of study drugs to death due to any cause over a period of 18 months.
Time to central nervous system (CNS) progression | Up to 1 year
  CNS progression will be defined as development of new CNS lesions detected on Brain MRI or CT scan, or in cerebrospinal fluid (CSF).
Peak plasma concentration (Cmax) of ceritinib + trametinib | Up to 1 year
  Measure peak plasma concentration (Cmax) of combination treatment ceritinib + trametinib

CONTACTS AND LOCATIONS:
Overall Officials: Collin Blakely, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Davis, Davis, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Derived] Lara MS, Gubens MA, Bacaltos B, Daran L, Lim SL, Li T, Gandara DR, Bivona TG, Riess JW, Blakely CM. Phase 1 Study of Ceritinib Combined With Trametinib in Patients With Advanced ALK- or ROS1-Positive NSCLC. JTO Clin Res Rep. 2022 Nov 21;3(12):100436. doi: 10.1016/j.jtocrr.2022.100436. eCollection 2022 Dec. PMID 36545322